CLINICAL TRIAL: NCT03972163
Title: Standardized PatiEnt-CenTered medicatiOn Review (SPECTORx) in Home Hospice
Brief Title: Standardized Patient-Centered Medication Review in Home Hospice
Acronym: SPECTORx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Utah (Other); Boston College (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer Tjia, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H00015417; 1R21AG060017 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-06-03 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hospices; Poly Pharmacy; Deprescriptions; Caregivers; Palliative Care; Prescription Drug Overuse; Interdisciplinary Communication
MeSH Terms: conditions — Prescription Drug Overuse

STUDY DESIGN:
Intervention Model Description: The Investigators will compare outcomes within and across 2 large hospice agencies using a cluster randomized trial study design.
Who Masked: Participant
Masking Description: Randomization to the educational intervention targeting hospice clinicians is at the level of the hospice. Within each of the 2 hospice agencies, The Investigators will randomize 1 office to intervention and 1 to control status. Outcomes assessment is at the level of the patient and family caregiver who will be masked to randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPECTORx Educational Intervention (Experimental): The program intervention is based on a combination of 3 existing, complementary, educational programs that, together, equip hospice staff to create a comprehensive, patient-centered, medication management care plan.
  Interventions: Behavioral: STOPPFrail (Screening Tool of Older Persons Prescriptions); Behavioral: "Discontinuing Medication Appropriately" and "Understanding the Art of Communication about Deprescribing"; Behavioral: "Key Approaches to Support Informal Family Caregivers in Managing Medications"
- Attention Control (Active Comparator): As the attention control, we will refer staff in control offices to the National Institute of Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Care Giver (FCG) support.
  Interventions: Behavioral: NIA Medication Management - Active Comparator

INTERVENTIONS:
Behavioral: NIA Medication Management - Active Comparator — As the attention control, we will refer staff in control offices to the National Institution on Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Care Giver (FCG) support.
  Arms: Attention Control
Behavioral: STOPPFrail (Screening Tool of Older Persons Prescriptions) — A screening tool used by clinicians with frail older adults with life-limiting illness to review medications
  Arms: SPECTORx Educational Intervention
Behavioral: "Discontinuing Medication Appropriately" and "Understanding the Art of Communication about Deprescribing" — Education resoruce used by clinicians to simplify and align medications with goals of care
  Arms: SPECTORx Educational Intervention
Behavioral: "Key Approaches to Support Informal Family Caregivers in Managing Medications" — Education resource used by clinicians to support Family Care Givers (FCGs)
  Arms: SPECTORx Educational Intervention

SUMMARY:
This is a pilot cluster randomized trial that tests the effect of a novel intervention that trains hospice staff to 1. regularly review, simplify, and align patients' prescribed medications with their goals of care as their illness progresses, and 2. support family caregivers with education that empowers them to understand each medication's use, develop skills for safe administration, and 3. understand when stopping medications may be beneficial.

DETAILED DESCRIPTION:
A tremendous challenge in home hospice care is ensuring that medication prescribing is appropriately aligned to patients' goals of care and that medications are appropriately managed by family caregivers. Therefore, the Investigators propose a novel intervention that trains hospice staff to 1. regularly review, simplify, and align patients' prescribed medications with their goals of care as their illness progresses, and 2. support family caregivers with education that empowers them to understand each medication's use, develop skills for safe administration, and understand when stopping medications may be beneficial. This program is called Standardized PatiEnt-CenTered medicatiOn Review (SPECTORx) in Home Hospice, and is based on a combination of 3 existing, complementary, educational programs that, together, train hospice staff to create a comprehensive, patient-centered, medication management care plan. The program also creates an online learning community that promotes ongoing education and practice change for hospice clinicians. This pilot study aims to demonstrate the feasibility of conducting a clinical trial to evaluate the efficacy of SPECTORx. The long-term objective is to test the hypothesis that SPECTORx reduces inappropriate medication prescribing and improves family caregiver reported quality of care. However, to accomplish this, the Investigators must first address challenging questions regarding the design, feasibility, and execution of trials in home hospice. The Investigators will accomplish this using a stakeholder engagement process to refine the SPECTORx intervention and trial protocol. The Investigators will then conduct a pilot cluster randomized trial and compare outcomes within and across 2 large, multi-office, hospice agencies from Utah and Massachusetts. Within each hospice agency, the Investigators will randomize 1 office to intervention and 1 office to attention control. Target enrollment is n=60 family caregiver-patient dyads of patients aged ≥65 years with advanced, life-limiting illness. Primary outcomes are acceptability and feasibility of the SPECTORx intervention by hospice stakeholders, and acceptability, burden and completion of family caregiver assessments (Family Caregiver Medication Administration Hassle Scale at baseline, 2 weeks, 4 weeks, 12 weeks, and quarterly). The overarching goal of this research is to align patient's prescribed medications with their goals of care at each stage of their advanced illness and to support family caregivers' medication management challenges. Ultimately, the Investigators want to improve the quality of medication prescribing, reduce treatment complexity and medication-related harm, and improve family caregiver outcomes for the almost 600,000 elderly Americans who receive home hospice services annually.

ELIGIBILITY:
Inclusion Criteria:

Patient - Newly admitted home hospice enrollees, aged ≥65 years old with:

* 1. advanced life-limiting illness;
* 2. an estimated life expectancy of >1 month;
* 3. recent functional status decline (defined as change in Karnofsky Performance Status [KPS] to < 80% in prior 3 months);
* 4. polypharmacy (defined as ≥ 5 regularly scheduled medications [excluding antimicrobials]);
* 5. cognitive ability to provide informed consent based on a Short Portable Mental Status Questionnaire (SPMSQ) score ≥6 OR, with a legally authorized representative who is willing and able to provide proxy consent.

Family ("any relative, partner, friend or neighbor who has a significant personal relationship with, and provides a broad range of assistance) Caregiver -

* self-identification as "usually" or "always" providing care to the eligible patient;
* English-speaking;
* telephone access; and
* cognitive ability to participate.

Exclusion Criteria:

Patient:

* Imminent death;
* pain crisis;
* no family caregiver or health care proxy

Family Caregiver:

* no telephone access;
* cognitive impairment.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tjia, MD, MSCE, Principal Investigator — UMass Medical School
Locations (1):
- Care Dimensions, Danvers, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tjia J, Clayton M, Chiriboga G, Staples B, Puerto G, Rappaport L, DeSanto-Madeya S. Stakeholder-engaged process for refining the design of a clinical trial in home hospice. BMC Med Res Methodol. 2021 Apr 30;21(1):92. doi: 10.1186/s12874-021-01275-0. PMID 33941089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at two hospice organizations where each hospice organization randomized 1 office to intervention and 1 office to control
Units Other Than Participants: hospice offices within hospice organizat
Period: Overall Study
Arm/Group | SPECTORx Educational Intervention | Attention Control
Started (Both Hospices) | 7; 2 hospice offices within hospice organizat (participants are patient-caregiver dyads) | 16; 2 hospice offices within hospice organizat (participants is number of patient-caregiver dyads)
Hospice 1 (units for cluster randomzed trial) | 5; 1 hospice offices within hospice organizat (participants is number of patient-caregiver dyads) | 12; 1 hospice offices within hospice organizat (participants is number of patient-caregiver dyads)
Hospice 2 (units for cluster randomized trial) | 2; 1 hospice offices within hospice organizat | 4; 1 hospice offices within hospice organizat
Completed (completed is for all dyad participants across both hospices) | 7; 2 hospice offices within hospice organizat (participants is number of patient-caregiver dyads in Hospice 1) | 15; 2 hospice offices within hospice organizat (participants is number of patient-caregiver dyads in Hospice 1)
Not Completed | 0; 0 hospice offices within hospice organizat | 1; 0 hospice offices within hospice organizat
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients: SPECTORx Educational Intervention; Caregivers SPECTORx Educational Intervention: The program intervention is based on a combination of 3 existing, complementary, educational programs that, together, equip hospice staff to create a comprehensive, patient-centered, medication management care plan.
  STOPPFrail (Screening Tool of Older Persons Prescriptions): A screening tool used by clinicians with frail older adults with life-limiting illness to review medications
  "Discontinuing Medication Appropriately" and "Understanding the Art of Communication about Deprescribing": Education resoruce used by clinicians to simplify and align medications with goals of care
  "Key Approaches to Support Informal Family Caregivers in Managing Medications": Education resource used by clinicians to support Family Care Givers (FCGs)
- Patients: Attention Control; Caregivers: Attention Control: As the attention control, we will refer staff in control offices to the National Institute of Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Care Giver (FCG) support.
  NIA Medication Management - Active Comparator: As the attention control, we will refer staff in control offices to the National Institution on Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Care Giver (FCG) support.
- Total: Total of all reporting groups
Arm/Group | Patients: SPECTORx Educational Intervention | Patients: Attention Control | Caregivers SPECTORx Educational Intervention | Caregivers: Attention Control | Total
Number analyzed (Participants) | 7 | 15 | 7 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants] — Population: Demographic data for Caregiver Intervention group missing/not available for select participants
  Participants
    number analyzed (Participants) | 7 | 15 | 6 | 15 | 43
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 3 | 8 | 11
    >=65 years | 7 | 15 | 3 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data for Caregiver Intervention group missing/not available.
  years
    number analyzed (Participants) | 7 | 15 | 0 | 0 | 22
    (all) | 83.6 (14.5) | 79.5 (10.3) |  |  | 80.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic data for Caregiver Intervention group missing/not available for select participants
  Participants
    number analyzed (Participants) | 7 | 15 | 6 | 15 | 43
    Female | 4 | 11 | 4 | 13 | 32
    Male | 3 | 4 | 2 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 7 | 14 | 6 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 6 | 13 | 5 | 13 | 37
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 15 | 7 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intervention Training Completion by Hospice Staff
Description: Number of Completed Intervention Trainings
Time Frame: Baseline
Population: Control group did not offer intervention training.
Measure: Count of Participants; unit: Participants
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 17 | 0
Participants | 17 | 0

2. Primary Outcome: Patient and Family Caregiver Eligibility Screens
Description: Number of Eligible Dyad Participants (i.e. participant = 1 dyad) screened for potential eligibility to inform subsequent eligibility criteria to obtain a sufficient study population.
Time Frame: 2 weeks prior to enrollment
Population: Screened dyads who met eligibility criteria
Measure: Number; unit: Dyads
Units Other Than Participants: Dyads
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 154 | 368
Number analyzed (Dyads) | 77 | 184
Dyads | 77 | 184

3. Primary Outcome: Patient and Family Caregiver Enrollment
Description: Number of Patients and Family Caregivers who enrolled
Time Frame: Baseline
Population: number of participants who consented to enrollment and survived to data collection; 1 patient died before data collection so dyad was removed
Measure: Number; unit: Dyads
Units Other Than Participants: Dyads
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 14 | 30
Number analyzed (Dyads) | 7 | 15
Dyads | 7 | 15

4. Primary Outcome: Completion of Primary Patient Outcome--Retention
Description: Number of Dyads who completed the Medication Regimen Complexity Score at Baseline
Time Frame: Baseline
Population: as for outcome 3
Measure: Number; unit: Dyads
Units Other Than Participants: Dyads
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 14 | 30
Number analyzed (Dyads) | 7 | 15
Dyads | 7 | 15

5. Secondary Outcome: Family Caregiver Medication Administration Hassle Scale
Description: The 24-item Family Caregiver Medication Administration Hassle Scale has four subscales: Information Seeking/Sharing, Safety Issues, Scheduling Logistics, and Polypharmacy. The theoretical range of the scores across 4 subscales is 0 to 120. Higher scores indicate greater burden. Overall scale reliability is .95.
Time Frame: Baseline, 2, 4, 6, 8 12, 16, 20, 24 weeks(or death)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 7 | 15
score on a scale
  Baseline | 13.6 (21.1) | 31 (16.7)
  2 weeks: number analyzed (Participants) | 3 | 11
  2 weeks | 19.7 (30.6) | 37 (17.5)
  4 weeks: number analyzed (Participants) | 3 | 9
  4 weeks | 16.7 (19.5) | 36.1 (17.5)
  6 weeks: number analyzed (Participants) | 2 | 5
  6 weeks | 22.5 (13.4) | 26.8 (12.2)
  8 weeks: number analyzed (Participants) | 2 | 4
  8 weeks | 21.5 (23.3) | 26.5 (9.5)
  12 weeks: number analyzed (Participants) | 1 | 4
  12 weeks | 10 | 33.3 (3.9)
  16 weeks: number analyzed (Participants) | 1 | 1
  16 weeks | 7 | 30
  20 weeks: number analyzed (Participants) | 0 | 1
  20 weeks |  | 47
  24 weeks (or death): number analyzed (Participants) | 0 | 1
  24 weeks (or death) |  | 21

6. Secondary Outcome: Medication Regimen Complexity Index
Description: Medication Regimen Complexity Index (MCRI) will characterize patients' chronic disease and preventive medication regimens (i.e. drugs initiated prior to hospice admission, not End of Life (EOL) symptom medications [e.g. haloperidol] because these increase over time). MRCI score weights dosage form, dosing frequency and administration instructions. Minimum MRCI is 1.5 [a single tablet once a day] and maximum score increases with medication number. Higher scores indicate greater complexity. MRCI score of 0 indicates no medication use. There is no established maximum score.
Time Frame: Baseline, 2, 4, 6, 8, 12, 16, 20, 24 weeks(or death)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 7 | 15
score on a scale
  baseline | 39 (8.8) | 23.5 (8.2)
  2 weeks: number analyzed (Participants) | 6 | 15
  2 weeks | 43.5 (13.1) | 31.0 (10.3)
  4 weeks: number analyzed (Participants) | 6 | 15
  4 weeks | 43.3 (12.9) | 32.5 (11.2)
  6 weeks: number analyzed (Participants) | 6 | 13
  6 weeks | 46.4 (13.9) | 33.6 (12.8)
  8 weeks: number analyzed (Participants) | 6 | 12
  8 weeks | 44 (19.4) | 31.1 (12.4)
  12 weeks: number analyzed (Participants) | 6 | 8
  12 weeks | 43.8 (21.1) | 26.8 (12.5)
  16 weeks: number analyzed (Participants) | 5 | 5
  16 weeks | 51.1 (11.3) | 29 (15.2)
  20 weeks: number analyzed (Participants) | 5 | 5
  20 weeks | 52.3 (12.3) | 33.4 (15.0)
  24 weeks (or death): number analyzed (Participants) | 4 | 5
  24 weeks (or death) | 47 (16.9) | 23.5 (22.6)

7. Secondary Outcome: Potential Adverse Event
Description: Hospitalizations and Emergency Department (ED) visits will be abstracted from the hospice record. Potential Adverse Drug Event (ADE)s and Adverse Drug Withdrawal Events (ADWEs) will be determined from medical record review
Time Frame: Week 2, 4, 6, 8, 12, 16, 20, 24
Population: Data on Potential Adverse Drug Events for patient participants
Measure: Number; unit: Adverse Events
Arm/Group | SPECTORx Educational Intervention | Attention Control
Number analyzed (Participants) | 7 | 15
Adverse Events
  Baseline | 0 | 0
  Week 2: number analyzed (Participants) | 6 | 15
  Week 2 | 0 | 0
  Week 4: number analyzed (Participants) | 6 | 15
  Week 4 | 0 | 0
  Week 6: number analyzed (Participants) | 6 | 13
  Week 6 | 0 | 0
  week 8: number analyzed (Participants) | 6 | 12
  week 8 | 0 | 0
  Week 12: number analyzed (Participants) | 6 | 8
  Week 12 | 0 | 0
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 0 | 0
  Week 20: number analyzed (Participants) | 5 | 5
  Week 20 | 0 | 0
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE were measured up to 24 weeks (or death)
Description: Any event due to the presence or progression of illness that a patient had on study enrollment are not be considered an adverse event (AE), since death more likely related to disease progression than not related to disease progression. Only events more likely not related to known underlying illness are considered an AE.
  Family caregivers were not assessed for All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events.
Groups:
- Patients: Attention Control: As the attention control, we will refer staff in control offices to the National Institute of Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Caregiver (FCG) support.
  NIA Medication Management - Active Comparator: As the attention control, we will refer staff in control offices to the National Institution on Aging (NIA)'s website on "Medicines and Medication Management" to review content and materials for use in Family Caregiver (FCG) support.
- Family Caregivers: SPECTORx Educational Intervention: Refer to "Patients: SPECTORx Educational Intervention" for description of intervention
- Family Caregivers: Attention Control: Refer to "Patients: Attention Control" for description of control
Arm/Group | Patients: SPECTORx Educational Intervention | Patients: Attention Control | Family Caregivers: SPECTORx Educational Intervention | Family Caregivers: Attention Control
All-Cause Mortality (participants affected / at risk) | 2/7 | 10/15 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/15 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/15 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT03972163/Prot_SAP_000.pdf